CLINICAL TRIAL: NCT06822855
Title: Changing Paragidms In The Prognostic Assessment Of Hodgkin Lymphoma
Acronym: LH_BIO
Status: Recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 696/2021/TESS/IRCCSRE
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-02

CONDITIONS: Classical Hodgkin Lymphoma; Classical Hodgkin Lymphoma Recurrent; Classical Hodgkin Lymphoma Refractory
Keywords: Liquid Biopsy; classical Hodgkin Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The mutational profile for Court A and Court B is defined through liquid biopsy, by analyzing DNA extracted from the patients' plasma. The DNA obtained from plasma is fully sequenced. For each patient, a peripheral blood sample is also collected, from which leukocytes are isolated and then control DNA is extracted. This sample of DNA is considered as free from disease and sequenced to exclude germline mutations not related to the tumor. Additionally, for Court A, a DNA sample is also extracted from FFPE material related to the diagnostic biopsy. This is done to verify that the mutational profile detected in the plasma recapitulates that obtained from the tumor biopsy. As for Court C, it consists of FFPE samples from which RNA is extracted and stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Post-Treatment Follow-Up Cohort (Cohort A): cHL patients who have completed active treatment and entered follow-up.
- Relapsed/Progressive Disease Cohort (Cohort B): cHL patients with a histological confirmation of relapse or disease progression.
- Retrospective cHL Cohort (Cohort C): Consecutive cHL patients from the archives of the Hematology Unit of AUSL-IRCCS, diagnosed between 2004 and 2019 and 250 cHL patients diagnosed between 2016 and 2021 from other Italian hematology centers.

SUMMARY:
Classical Hodgkin's Lymphoma (cHL) is a rare but highly treatable malignancy of the immune system, primarily affecting young adults. Despite significant therapeutic advancements, frontline treatment failure occurs in up to 30% of cases, with relapse or refractory disease affecting over 50% of these patients. The main therapeutic challenge in cHL remains achieving an optimal balance between disease control and reducing long-term adverse effects. Current prognostic tools only partially capture patient heterogeneity, and cHL continues to evolve spatially and temporally throughout the course of the disease. Personalized treatment strategies require novel integrated tools that better monitor tumor complexity and anticipate disease progression.

Fluorodeoxyglucose positron emission tomography (FDG-PET) has improved risk stratification in cHL, as metabolic response during or after chemotherapy strongly correlates with disease progression and survival. However, FDG-PET has limitations, including the absence of standardized criteria and the necessity to initiate treatment before response assessment. To overcome these limitations, molecular profiling and radiomic analysis of baseline FDG-PET data may provide deeper insights into tumor biology, improving prognostic accuracy.

This observational study aims to dissect the genetic and phenotypic heterogeneity of cHL at diagnosis and during disease evolution, with the goal of identifying novel prognostic biomarkers. These findings could lead to better treatment personalization, increasing cure rates while minimizing treatment-related toxicity. The study is based on the hypothesis that correlating DNA profiling at diagnosis, gene expression, and radiomic features may enable the identification of high-risk signatures, refining prognostic models in cHL. Additionally, liquid biopsy represents a non-invasive method for assessing tumor mutational complexity. The analysis of circulating DNA (cDNA) throughout disease progression could provide insights into genetic evolution and help predict overt progression before clinical manifestations occur.

The primary objective is to define the genetic mutational profile of cHL at disease progression. As secondary objectives, it will evaluate whether liquid biopsy can accurately recapitulate the genetic heterogeneity observed in tumor tissue, determine the predictive accuracy of liquid biopsy in anticipating disease progression, and correlate genomic and radiomic features with patient outcomes to refine risk stratification and therapeutic decision-making.

By integrating molecular and imaging-based biomarkers, this study aims to enhance personalized treatment strategies, improve risk-adapted therapeutic approaches, and ultimately optimize curability and quality of life for patients with cHL.

DETAILED DESCRIPTION:
This study has both retrospective and prospective components. The prospective part includes patients with Classical Hodgkin's Lymphoma (cHL) who have completed active treatment and entered follow-up (Cohort A), as well as patients with a histological confirmation of relapse or progression (Cohort B). The retrospective cohort (Cohort C) consists of 235 consecutive cHL patients collected from the archives of the Hematology Unit of AUSL-IRCCS between 2004 and 2019, along with up to 250 cHL patients diagnosed between 2016 and 2021 from other Italian hematology centers.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 anni
* Written informed consent signed

Cohort A

* Age >18 years
* Histologically confirmed diagnosis of relapsed/refractory classical Hodgkin lymphoma identified during induction or follow-up
* Available formalin-fixed, paraffin-embedded (FFPE) biopsy at diagnosis and at the time of progression/relapse
* Available plasma sample at progression (before the beginning of salvage therapy)
* Available FDG-PET evaluation at study enrollment
* Available clinical, laboratory, and radiologic data at diagnosis and relapse

Cohort B

* Diagnosis of classical Hodgkin lymphoma
* Completion of first-line standard systemic treatment (chemotherapy-based or chemoradiotherapy combined modality)
* Available plasma sample at the end of treatment (at least 30 days from the last chemotherapy)
* Available FFPE biopsy at diagnosis
* No further treatment planned
* Available clinical, laboratory, and radiologic data at diagnosis and response evaluation
* Patient's willingness to undergo 6 months follow-up plasma sample collection and to attend regular follow-up

Cohort C

* Histologically confirmed diagnosis of classical Hodgkin lymphoma
* Standard treatment as per available guidelines (e.g., ESMO guidelines)
* Available treatment data, response, and follow-up data
* Available FFPE biopsy at diagnosis
* Available FDG-PET evaluation at study enrollment

Exclusion Criteria:

* Patients with nodular lymphocyte predominant Hodgkin lymphoma are not eligible; all other subtypes including nodular sclerosis, lymphocyte-depleted, lymphocyte-rich, and mixed cellularity Hodgkin lymphoma may be enrolled.
* Active HIV, HBV, HCV viral infection
* Concomitant neoplasm not treated with a curative aim

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will involve three patient cohorts, with participants recruited from multiple centers across Italy during routine follow-up visits.
  Cohort A will include 70 patients with classical Hodgkin lymphoma (cHL) who have a histological confirmation of relapse or progression. These patients will be enrolled at the time of disease relapse/progression, and plasma samples for ctDNA analysis will be collected concurrently.
  Cohort B will consist of 200 cHL patients who have completed active treatment and entered the follow-up phase. Plasma samples will be collected from these patients at the time of enrollment (P0) and again at a six-month follow-up (P6FU). This cohort will be followed for a minimum of two years from the time of enrollment.
  Cohort C is a retrospective cohort that will be divided into two subgroups:
  Training cohort: 235 consecutive cHL patients collected from the archives of the Hematology Unit of AUSL-IRCCS between 2004 and 2019. This cohort is representative of the ge
Sampling Method: Non-Probability Sample
Enrollment: 755 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Genetic Mutational Profiling of cHL at Progression | At enrollement
  The mutational profile of Classical Hodgkin's Lymphoma patients enrolled in Cohort A will be generated using deep sequencing technologies, including Cancer Personalized Profiling by deep-sequencing (CAPP-seq), on biopsy samples collected at the time of initial diagnosis and at the time of progression to identify key alterations associated with disease progression and aggressiveness.

SECONDARY OUTCOMES:
Liquid Biopsy Ability to Recapitulate Tissue Genetic Heterogeneity | Up to 4 years
  Circulating tumor DNA (ctDNA) from plasma samples collected at baseline (Cohort B) and at the time of disease progression (Cohorts A and B) will be analyzed using CAPP-seq and compared with matched germline DNA (gDNA). Identified mutations will be compared to a background variant database to filter out technical sequencing errors and identify true positive alterations. Heatmaps and COSMIC database annotations will be used to assess the functional relevance of selected variants. The mutational profile in plasma will be compared with biopsy results obtained at progression to evaluate the ability of ctDNA to capture tumor heterogeneity and progression-related alterations.
Accuracy of Liquid Biopsy in Anticipating Disease Progression | From 2 up to 4 years
  Plasma samples of Cohort B patients will be collected at enrollement and at 6 months of follow-up, and the presence of mutations will be assessed using deep sequencing (CAPP-seq). The results will be compared with clinical outcomes over a follow-up period of at least 2 years to determine the specificity and sensitivity of liquid biopsy in predicting progression.
Correlation between Gene Expression Profiling and Progression-free survival (PFS) | Up to 4 years
  Gene expression profiling conducted on tissue samples from subjects in Cohort C at diagnosis will be correlated with progression-free survival (PFS).
Correlation between Gene Expression Profiling and cnical events like relapse and refractoriness | Up to 4 years
  Gene expression profiling conducted on tissue samples from subjects in Cohort C at diagnosis will be correlated with cnical events like relapse and refractoriness).

CONTACTS AND LOCATIONS:
Overall Officials: Luminari Stefano, MD, Principal Investigator — Azienda USL - IRCCS di Reggio Emilia
Locations (12):
- Italy (12):
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, RE
  - A.O.S.G. Moscati, Avellino
  - Spedali Civili Brescia, Brescia
  - Istituto Oncologico Veneto, Padua
  - Azienda Ospedaliera "Ospedali Riuniti Villa Sofia-Cervello", Palermo
  - Azienda Ospedaliera di Perugia, Perugia
  - Ospedale S. Maria della Misericordia, Azienda Ospedaliera di Perugia, Perugia
  - AUSL Piacenza, Piacenza
  - Azienda Ospedaliera Santa Maria - Terni, Terni
  - AOU Città della salute e della Scienza, "Le Molinette", Torino
  - AOU Città della Salute e della Scienza, Torino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Merli F, Luminari S, Gobbi PG, Cascavilla N, Mammi C, Ilariucci F, Stelitano C, Musso M, Baldini L, Galimberti S, Angrilli F, Polimeno G, Scalzulli PR, Ferrari A, Marcheselli L, Federico M. Long-Term Results of the HD2000 Trial Comparing ABVD Versus BEACOPP Versus COPP-EBV-CAD in Untreated Patients With Advanced Hodgkin Lymphoma: A Study by Fondazione Italiana Linfomi. J Clin Oncol. 2016 Apr 10;34(11):1175-81. doi: 10.1200/JCO.2015.62.4817. Epub 2015 Dec 28. PMID 26712220
- [Background] Andre MPE, Girinsky T, Federico M, Reman O, Fortpied C, Gotti M, Casasnovas O, Brice P, van der Maazen R, Re A, Edeline V, Ferme C, van Imhoff G, Merli F, Bouabdallah R, Sebban C, Specht L, Stamatoullas A, Delarue R, Fiaccadori V, Bellei M, Raveloarivahy T, Versari A, Hutchings M, Meignan M, Raemaekers J. Early Positron Emission Tomography Response-Adapted Treatment in Stage I and II Hodgkin Lymphoma: Final Results of the Randomized EORTC/LYSA/FIL H10 Trial. J Clin Oncol. 2017 Jun 1;35(16):1786-1794. doi: 10.1200/JCO.2016.68.6394. Epub 2017 Mar 14. PMID 28291393
- [Background] Eichenauer DA, Aleman BMP, Andre M, Federico M, Hutchings M, Illidge T, Engert A, Ladetto M; ESMO Guidelines Committee. Hodgkin lymphoma: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2018 Oct 1;29(Suppl 4):iv19-iv29. doi: 10.1093/annonc/mdy080. No abstract available. PMID 29796651
- [Background] Hoppe RT, Advani RH, Ai WZ, Ambinder RF, Aoun P, Armand P, Bello CM, Benitez CM, Bierman PJ, Chen R, Dabaja B, Dean R, Forero A, Gordon LI, Hernandez-Ilizaliturri FJ, Hochberg EP, Huang J, Johnston PB, Kaminski MS, Kenkre VP, Khan N, Maddocks K, Maloney DG, Metzger M, Moore JO, Morgan D, Moskowitz CH, Mulroney C, Rabinovitch R, Seropian S, Tao R, Winter JN, Yahalom J, Burns JL, Ogba N. NCCN Guidelines Insights: Hodgkin Lymphoma, Version 1.2018. J Natl Compr Canc Netw. 2018 Mar;16(3):245-254. doi: 10.6004/jnccn.2018.0013. PMID 29523663
- [Background] Luminari S, Donati B, Casali M, Valli R, Santi R, Puccini B, Kovalchuk S, Ruffini A, Fama A, Berti V, Fragliasso V, Zanelli M, Vergoni F, Versari A, Rigacci L, Merli F, Ciarrocchi A. A Gene Expression-based Model to Predict Metabolic Response After Two Courses of ABVD in Hodgkin Lymphoma Patients. Clin Cancer Res. 2020 Jan 15;26(2):373-383. doi: 10.1158/1078-0432.CCR-19-2356. Epub 2019 Oct 23. PMID 31645353
- [Background] Rossi D, Spina V, Bruscaggin A, Gaidano G. Liquid biopsy in lymphoma. Haematologica. 2019 Apr;104(4):648-652. doi: 10.3324/haematol.2018.206177. Epub 2019 Mar 7. No abstract available. PMID 30846503
- [Background] Spina V, Bruscaggin A, Cuccaro A, Martini M, Di Trani M, Forestieri G, Manzoni M, Condoluci A, Arribas A, Terzi-Di-Bergamo L, Locatelli SL, Cupelli E, Ceriani L, Moccia AA, Stathis A, Nassi L, Deambrogi C, Diop F, Guidetti F, Cocomazzi A, Annunziata S, Rufini V, Giordano A, Neri A, Boldorini R, Gerber B, Bertoni F, Ghielmini M, Stussi G, Santoro A, Cavalli F, Zucca E, Larocca LM, Gaidano G, Hohaus S, Carlo-Stella C, Rossi D. Circulating tumor DNA reveals genetics, clonal evolution, and residual disease in classical Hodgkin lymphoma. Blood. 2018 May 31;131(22):2413-2425. doi: 10.1182/blood-2017-11-812073. Epub 2018 Feb 15. PMID 29449275